CLINICAL TRIAL: NCT06163937
Title: Examining the Acute Effects of Two Different Fruit Juices (Orange Juice and Mixed Fruit Juice Consisted of Apple, Orange, Grape, and Pomegranate) on Postprandial Glycemic Responses and Satiety in Healthy Individuals
Brief Title: Acute Effects of Fruit Juices Consumption on Postprandial Glycemic Responses and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Collaborators: Institute of Technology and Agricultural Products (Unknown)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: HRBD 67/06.09.2023
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetitive Behavior
Keywords: blood glucose; fruit juice; glycemic index; glycemic load; satiety
MeSH Terms: conditions — Appetitive Behavior | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glucose as reference food (Experimental): Ten healthy, normal-weight adults after 10-14 hours of fasting, consumed 50g available carbohydrates from D-glucose, tested three times, in different visits as reference food; and 50g available carbohydrates from orange juice and mixed fruit juice (consisted of apple, orange, grape, and pomegranate), each tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after beverage consumption. The first glucose sample was taken exactly 15min after the first sip of drink.
  Interventions: Other: Glucose as reference food
- Orange juice (Experimental): Ten healthy, normal-weight adults after 10-14 hours of fasting, consumed 50g available carbohydrates from D-glucose, tested three times, in different visits as reference food; and 50g available carbohydrates from orange juice and mixed fruit juice (consisted of apple, orange, grape, and pomegranate), each tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after beverage consumption. The first glucose sample was taken exactly 15min after the first sip of drink.
  Interventions: Other: Orange juice
- Mixed fruit juice (Experimental): Ten healthy, normal-weight adults after 10-14 hours of fasting, consumed 50g available carbohydrates from D-glucose, tested three times, in different visits as reference food; and 50g available carbohydrates from orange juice and mixed fruit juice (consisted of apple, orange, grape, and pomegranate), each tested once, in different visits, along with 300mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min after beverage consumption. The first glucose sample was taken exactly 15min after the first sip of drink.
  Interventions: Other: Mixed fruit juice

INTERVENTIONS:
Other: Glucose as reference food — Ten healthy, normal-weight subjects after 10-14 hours of fasting, consumed 50g glucose diluted in 300ml water, tested three times, in different visits, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
  Arms: Glucose as reference food
Other: Orange juice — Ten healthy, normal-weight subjects after 10-14 hours of fasting, consumed 50g available carbohydrates from orange juice, tested once, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
  Arms: Orange juice
Other: Mixed fruit juice — Ten healthy, normal-weight subjects after 10-14 hours of fasting, consumed 50g available carbohydrates from mixed fruit juice (consisted of apple, orange, grape, and pomegranate), tested once, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
  Arms: Mixed fruit juice

SUMMARY:
This study investigated the acute effects of two fruit juices on postprandial glycemic responses and satiety in healthy individuals

DETAILED DESCRIPTION:
This study aimed to 1. Determine the glycemic index and glycemic load of two types of fruit juices (orange juice and mixed fruit juice consisted of apple, orange, grape, and pomegranate) and 2. Investigate the effects of these two fruit juices on postprandial glycemic responses and satiety in healthy individuals

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking
* non-diabetic and normotensive men and women
* body mass index between 18.5 and 25 kg/m2

Exclusion Criteria:

* severe chronic disease (e.g. cardiovascular diseases, diabetes mellitus, kidney or liver conditions, endocrine conditions)
* gastrointestinal disorders
* pregnancy
* lactation
* competitive sports
* alcohol abuse
* drug dependency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Glycemic index | 2 hours
  Glucose solution (50 g) was the reference food (GI = 100%) against which all test foods were compared. Subjects arrived at the laboratory at eight to nine o'clock in the morning after 10-12 h overnight fast. Each subject was fed equivalent 50 g available carbohydrate of test foods or reference food in random order. To minimize day to day variation of glucose tolerance, the reference food was tested in triplicate in each subject. All test and reference foods were served with 250 mL of water. An automatic lancet device and glucometer (calibrated MediSmart Ruby glucose meter with a lancing device, Lilly-PHARMASERV SA, Greece) was used for finger capillary blood samples. Blood samples were taken immediately before the start of the study (0 min) and 15, 30, 45, 60, 90 and 120 min after the start of eating.
Capillary blood glucose responses | 2 hours
  Clinically useful change in blood glucose, defined as the restoration of glucose within normal limits during the 2hr glucose tolerance test

SECONDARY OUTCOMES:
Subjective appetite ratings | 2 hours
  Useful change in subjective appetite using visual analogue scales with a score 0 to 10 (given in the form of booklet, one scale per page) at baseline, 15, 30, 45, 60, 90 and 120min. The minimum or maximum score will be evaluated if it is better or worse depending on the appetite variable e.g. hunger, satiety, desire to eat, etc.
Blood pressure | 2 hours
  Useful change in systolic and diastolic blood pressure 2 hours post-consumption of tested beverages

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (2):
- Greece (2):
  - Agricultural University of Athens, Athens, Attica
  - Agricultural University of Athens, Athens

IPD SHARING:
Plan to Share IPD: No